CLINICAL TRIAL: NCT03515161
Title: Computer-assisted Vasopressor Infusion for Hemodynamic Optimization in Patients Undergoing High Risk Surgery
Brief Title: Closed-Loop Titration of Vasopressor Infusions: Feasibility Study or Proof of Concept Study
Acronym: CLV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, Principal Investigator, Erasme University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P2018/276
Record Dates: First submitted 2018-04-17; First posted 2018-05-03 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Closed-Loop Communication; Hemodynamic Instability
Keywords: closedloop; vasopressor
MeSH Terms: conditions — Teach-Back Communication

STUDY DESIGN:
Intervention Model Description: SINGLE GROUP ASSIGNMENT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Closed-loop (Experimental): Study patients will receive a baseline crystalloid infusion of 3 cc/kg/hr and all additional fluid management will be performed manually using the assisted fluid management sofware from the EV1000 monitor. A closed-loop system will automatically administer vasopressor based on the predefined target MAP chosen by the anesthesiologist in charge of the patient
  Interventions: Device: closed-loop

INTERVENTIONS:
Device: closed-loop — Vasopressor admnistration in the closed loop group will be performed via a closed loop (automated) system that will use an infusion pump (Q-Core) and a controller (a computer run index and algorithm developed by Sironis) to make frequent, regular and accurate adjustments to the amount of vasopressor the patient receives using feedback from standard operating room monitors.

SUMMARY:
The purpose of this study is to evaluate the performance of a novel closed-loop (automated) vasopressor administration system that delivers norepinephrine using feedback from standard operating room hemodynamic monitor (EV1000 Monitor-Flotrac or Clearsight system, Edwards Lifesciences, IRVINE, USA).

DETAILED DESCRIPTION:
In this protocol, the investigators will report the percentage of case time in hypotension (defined as Mean arterial pressure (MAP) < 65mmHg). The target MAP will be set at 70mmHg, except for neuro embolisation case where MAP can be higher. The investigators want to demonstrate that the closed-loop system can prevent hypotension at this specific set point.

The Investigators have shown this to be the case in simulation studies and in-vivo animal studies (under submission) but not yet experimentally in a clinical setting. Investigators will recruit their patients from the surgical record that that require a mini-invasive or a non-invasive cardiac output monitoring (EV1000 monitoring using the Flotrac or clearsight system) ; either high risk patients undergoing high risk surgery (vascular-cardiac- Major Abdominal or renal transplant, neuro-endo-vascular surgery (aneuvrysm) and require mechanical ventilation and consent to participate in the study will be included in the study.

The investigators will also test the system in a short series of patients in the ICU setting ( critically ill patients): ideally in 3-4 "types" of patients ( septic patients, neuro ICU patients, ARDS patients and postoperative patients( ideally intubated patients or sedated patients) .The target mean arterial pressure can be different from the 70 mmHg of the surgical patients especially for the neurologic patients (head trauma injury patients or neuro-endovascular surgical patients). In these two subgroups of patients, the target MAP can even vary during the case depending on the surgeons requests (neuro radiologists) or depending on cerebral autoregulation.

Participants will receive standard patient care in that in no way will their anesthetic or surgical procedure will be altered as part of the study, with the exception of vasopressor administration. Fluids will be given as goal directed therapy using the assisted fluid management software present in the EV1000 monitor (only for vascular and abdominal cases).

The closed loop (automated) system will use an infusion pump (Q-Core) and a controller (a computer run index and algorithm developed by Sironis) to make frequent, regular and accurate adjustments to the amount of vasopressor infusion rate the patient receives using feedback from standard operating room monitors at ERASME HOSPITAL Data from this study will also be retrospectively compared to subjects case matched to evaluate differences in MAP time in target, total amount of vasopressor received, and patient outcomes (for patients undergoing high risk surgery and/or neuro endovascular patients)

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 18
* Subjects undergoing elective high risk surgery (either vascular-cardiac- or transplant)
* Subjects requiring general anesthesia and mechanical ventilation
* Subjects requiring cardiac output monitoring with an arterial line

Exclusion Criteria:

* Subjects under 18 years of age
* Subjects not undergoing surgery
* Subjects not requiring general anesthesia or mechanical ventilation
* Subjects not requiring cardiac output monitoring or an arterial line
* Subject with Atrial Fibrillation
* Subjects who are pregnant
* Subjects without the capacity to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Percentage of case Time in hypotension (MAP <65 mmHg) for surgical patients. For potential recrutment of critically ill patients in the ICU, this target can be different (higher, depending on the type of patient and comorbidities) | At postoperative day 1
  The primary outcome will be the percentage of case time in predefined MAP target

SECONDARY OUTCOMES:
percentage of case time with MAP >75 mmHg with norepinephrine still running | At postoperative day 1
  overtreatment
Amount of vasopressors received | At postoperative day 1
  Amount of vasopressors received

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, M.D, Principal Investigator — Erasme
Locations (1):
- Erasme, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Yes
We can provide individual patients data ( all hemodynamic data)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the completion of the study and the publication of the results
Access Criteria: Contact PI

REFERENCES:
- [Derived] Joosten A, Alexander B, Duranteau J, Taccone FS, Creteur J, Vincent JL, Cannesson M, Rinehart J. Feasibility of closed-loop titration of norepinephrine infusion in patients undergoing moderate- and high-risk surgery. Br J Anaesth. 2019 Oct;123(4):430-438. doi: 10.1016/j.bja.2019.04.064. Epub 2019 Jun 27. PMID 31255290